CLINICAL TRIAL: NCT05285007
Title: Limited Ankle Dorsiflexion and Effect on Single Limb Squats in Individuals With Patellofemoral Pain: Interventions and Outcomes in a Randomized Clinical Trial
Brief Title: Limited Ankle Dorsiflexion and Effect on Single Limb Squats in Individuals With Patellofemoral Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5220026
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Movement; Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Intervention Group (Experimental): The experimental group will receive two interventions to increase dorsiflexion range of motion.
  Interventions: Other: Mobilization with Movement
- Minimal Intervention Group (Active Comparator): The minimal intervention group will read and infographic and complete 5 minutes of treadmill walking.
  Interventions: Other: No mobilization with movement and education

INTERVENTIONS:
Other: Mobilization with Movement — Participants will be lunging on a box with posterior ankle glide of 10 seconds times 5 sets. They will have 30 seconds rest between trials. Participant will have their ankle taped and then walk on a treadmill at a self-selected pace for 5 minutes.
  Arms: Primary Intervention Group
Other: No mobilization with movement and education — Participants ankle will not be taped and they will walk on the treadmill for 5 minutes and receive education.
  Arms: Minimal Intervention Group

SUMMARY:
The purpose of this graduate student research study is to investigate the relationship between limited ankle dorsiflexion and the potential effects on a single limb squat task in the Patellofemoral/Knee Pain population.

DETAILED DESCRIPTION:
1. Participants will undergo Covid screening prior to filling out consent form and PHI. Randomization will occur to create an experimental group and a minimal intervention group.
2. Participants will complete two self-reported questionnaires on how their diagnosis affects functional activities.
3. Dorsiflexion range of motion in a weight bearing position will be taken.
4. Hip abductor strength on tested limb will be measure on isokinetic device.
5. The Lateral Step Down test will be conducted for 6 trials on each participant, 3 with a heel wedge and 3 without, movement recorded, and graded using two motion capture devices.
6. The experimental group will receive two interventions to increase dorsiflexion range of motion. The minimal intervention group will read and infographic and complete 5 minutes of treadmill walking.
7. Each participant will then have their dorsiflexion measured again prior to completing another 3 trials of the Lateral Step Down test.

ELIGIBILITY:
Inclusion Criteria:

* History of active Patellofemoral Pain for at least 6 months
* No clinic based therapeutic interventions for a 6-month period prior to testing
* Females aged 18-59 years' old
* Limited ankle dorsiflexion as noted by <45degs using the weight bearing lunge test

Exclusion Criteria:

* History of musculoskeletal surgery or fractures on the tested leg or lumbar spine that could affect their biomechanics during the study
* History of soft tissue or skeletal abnormalities in the tested limb
* Current knee effusion
* Resting pain greater than 5/10

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Weight bearing lunge test | change between baseline and post intervention on Day 1
  This test is used to assess a participant's available dorsiflexion range of motion in a weight bearing position. Furthermore, this places the participants hip, knee, and ankle into a flexed position which correlates with the squat tests we will be using.

SECONDARY OUTCOMES:
Patellofemoral Disability Index | change between baseline and post intervention on Day 1
  The Index is a self-reported questionnaire that addresses the amount of pain a person may have during tasks such as running, jumping, and stair climbing.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, Dsc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States